CLINICAL TRIAL: NCT05054894
Title: Open Label Study for the Use of Plasmapheresis for Treatment of Age-Related Frailty
Brief Title: Plasmapheresis for Treatment of Age-Related Frailty
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PlasmapheresisFrailty2021
Record Dates: First submitted 2021-08-30; First posted 2021-09-23 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Age-Related Frailty
MeSH Terms: interventions — Plasma Exchange; Plasmapheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Plasmapheresis for Age-Related Frailty) (Experimental): Participants will receive plasmapheresis once a month for six months. All participants will be in this arm.
  Interventions: Other: Therapeutic Plasma Exchange (TPE)

INTERVENTIONS:
Other: Therapeutic Plasma Exchange (TPE) — Following all necessary screening and consenting protocol, patients will be scheduled for the plasmapheresis procedure.
  Plasmapheresis
  On the days of the scheduled procedure, patients will undergo up to 1.5 hours of plasmapheresis treatment. Patients will be awake and situated in a relaxed position in a reclined chair. The plasmapheresis device to be used is the Fresenius Kabi 'Amicus', which is currently FDA approved for a variety of clinical conditions. In one treatment, roughly 60-70% of a patient's plasma can safely be replaced; by using six consecutive treatments, more of the patient's plasma (approaching 100%) will be replaced in an exponential fashion.
  Other Names: Plasmapheresis

SUMMARY:
This study is designed to evaluate the efficacy of albumin-infused plasmapheresis, using the Fresenius Kabi 'Amicus' apheresis machine, among patients with age-related frailty characterized by reduced physical, cognitive and immunological functioning. Additionally, this study is designed to evaluate the safety and tolerability of repeated plasmapheresis treatment.

DETAILED DESCRIPTION:
As population aging continues to accelerate around the world, there is increasing recognition of health burdens related to frailty. Age-related frailty indisputably reduces quality of life for an aging-individual, as well as for caregiving individuals. To date, there is no proven effective therapy or cure for age-related frailty. There is an urgent need to address the burden of frailty with possible therapeutic solutions.

One model proposed nine hallmarks of aging which fall into three categories: 1) primary causes of cellular damage (e.g., genomic instability, telomere attrition, epigenetic alterations, loss of proteostasis); 2) compensatory or antagonistic responses to damage (e.g., deregulated nutrient sensing; mitochondrial dysfunction, cellular senescence); and 3) the integrative result of (1) and (2) that is considered responsible for functional decline (e.g., stem cell exhaustion, altered intercellular communication). In more recent reports, frailty has been defined as a syndrome related to the fatigue of physiological systems; in other words, it is "a state of increased vulnerability to poor resolution of homeostasis after a stressor event and is a consequence of cumulative decline in many physiological systems during a lifetime. This cumulative decline depletes homeostatic reserves until minor stressor events trigger disproportionate changes in health status". This definition of frailty as a syndrome whose incidence increases with aging is based on research that highlights its relationship with various biological processes rather than chronological age.

It has been proposed that an underlying mechanism leading to many frailty-related neurological diseases is a gradual build up of certain molecules in patients' plasma. Molecules such as auto-antibodies develop naturally over time in response to disease over a patient's life span, but build up of these molecules has been linked to both central and peripheral nervous system disorders such as Alzheimer's and Parkinsons. Specifically, beta-amyloid accumulation and toxic autoimmunity-related proteins have been used as markers of aging-related neurological diseases such as Alzheimer's Disease (AD) and multiple sclerosis (MS). Considering this, a successful treatment for many neurological disorders including those listed has been the process of Plasmapheresis. In Plasmapheresis, the process is to extract some of a patient's blood, remove a percentage of the plasma in the blood, and finally replace it with either 1) donor plasma, 2) albumin, or 3) a combination of saline with albumin. This process ultimately dilutes the amount of harmful molecules. The American Society for Apheresis (ASFA) has determined that Plasmapheresis is accepted as a Category 1 (or first-line therapy) for nervous system disorders that exhibit frailty symptoms such as: Acute Inflammatory Demyelinating Polyneuropathy (Guillain-Barre Syndrome), Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP), Multiple Sclerosis (MS), and more.

Studies have suggested low serum hypoalbuminemia (albumin) is a significant risk factor for frailty in elderly patients. Therefore, a possible treatment approach for age-related frailty is to not only remove the build up of harmful molecules with plasmapheresis, but to replenish serum albumin during reinfusion. A recent study demonstrated that utilizing albumin in plasmapheresis decreased concentration of Amyloid-Beta plaque build up in cerebrospinal fluid, as well as increased scores on cognitive, functional, and behavioral tests in elderly patients with Alzheimer's Disease. The present study is therefore designed to assess clinical benefit of plasmapheresis with albumin in patients with age related frailty.

Design

The present study is being undertaken as an open-label study to evaluate the safety and feasibility of plasmapheresis as an intervention for patients with age-related frailty. Baseline and outcome measures in this study utilize validated tests that are appropriate for repeated measures. The present study can be easily implemented because instruments have been in routine clinical deployment providing for a high degree of availability and reliability. Quality assurance is tightly controlled. The study population is sufficiently broad and the conditions of interest are sufficiently prevalent so that recruitment of subjects is not a limiting factor.

The safety of this protocol will be closely monitored and data will be used to determine whether any significant safety issues exist when using plasmapheresis. Adverse events will be noted whenever they occur but will be recorded at the time of the procedure and throughout routine follow-ups, which will persist weekly throughout the duration of the active study protocol.

All patients will have a thorough discussion to obtain informed consent. If the patient is unable to provide consent due to cognitive decline, consent will be provided by a legally authorized representative (LAR). Additional meetings with the physicians will further clarify the nature of the study and the possible risks involved. The nature of this study does not require randomization, but rather attempts to isolate adverse and advantageous events should they occur.

Patients deemed appropriate candidates for plasmapheresis will be treated for a total of 6 sessions; 1 session per week or month - This time frame is dependent on the acuteness of the patient's condition.. Each treatment will take roughly 1.5 hours to complete, depending on the specific patient's needs.

Subjects

The subjects in this research study will be recruited through medical practice. There are no enrollment restrictions based on race or ethnic origin. There are also no additional benefits, risks, advantages, or disadvantages based on any race or ethnic origin. This study will seek to enroll a total of 100 subjects.

ELIGIBILITY:
Inclusion: In order for a subject to be considered for the inclusion in this study, the following criteria are required:

* Age eligibility requirements fall in a range from 50 to 95 years of age
* Clinical appraisal by physician indicating signs of frailty (apart from a co-occurring condition), scoring 3<x <7 as denoted by the CSHA Clinical Frailty Scale (see Appendix A; Rockwood, Song, MacKnight, et al, 2005; Golpanian, DiFede, Pujol, et al., 2016)

Exclusion: In order for a subject to be considered for this study, he/she may NOT have any of the following

* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Pregnancy, women who may become pregnant or are breastfeeding
* Advanced terminal illness
* Subjects with rash or open wounds (for example from treatment of squamous cell cancer)
* Subjects with a reactive serologic test positive for Syphilis

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in Canadian Study of Health and Aging (CSHA) Clinical Frailty Scale | Change in Scale Score after completion of study (6 months)
  A global clinical measure of fitness and frailty in elderly people, ranging from 1-9, with 1 being 'Very Fit', and 9 being 'Terminally I'll'. Reduction in score from higher to lower is to be seen as improvement in frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, M.D., Principal Investigator — Neurological Associates The Interventional Group
Locations (1):
- Neurological Associates - The Interventional Group, Santa Monica, California, United States